

Ysbyty Athrofaol Cymru University Hospital of Wales



IRAS ID: 238464 Study ID Number:

Patient Identification Number:

## PARTICIPANT RE- CONSENT FORM 2 [Version 2.0 30/01/18]

| PARTICIPANT RE | E- CONSENT FORM 2 | [Version 2.0 30/01/1 | oj |
|---|---|---|---|
| Title of Study: Measuring Phys | sical Activity Levels in | Critical Care: A Feas | ibility Study |
| Name of Researchers: Mrs La | ura Jones, Dr Harriet S | | ease initial box |
| 1. I confirm that I have read and understand the information sheet dated 30/01/18 [version 2.0] for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | |
| 2. I understand that my participation at any time without giving any rebeing affected. | • | | |
| 3. I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from regulatory authorities, University College London or from Cardiff and Vale UHB, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | |
| 4. I agree for the data already colled device to be used for this resea | | ring the activPAL™ | |
| 5. I agree to take part in the abov | e study. | | |
| 6. I would like to receive a copy of the findings of the study: Yes No | | | No |
| Name of patient | Date | Signature | |
| Name of person taking consent | <br>Date | Signature | |